CLINICAL TRIAL: NCT04421820
Title: A Phase 1b/2a Dose Escalation Study of BOLD-100 in Combination With FOLFOX Chemotherapy in Patients With Advanced Solid Tumours
Brief Title: BOLD-100 in Combination With FOLFOX for the Treatment of Advanced Solid Tumours
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bold Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BOLD-100-001
Record Dates: First submitted 2020-05-26; First posted 2020-06-09 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer; Pancreatic Cancer; Gastric Cancers; Cholangiocarcinoma
MeSH Terms: conditions — Colorectal Neoplasms; Pancreatic Neoplasms; Stomach Neoplasms; Cholangiocarcinoma | interventions — Leucovorin; Fluorouracil; Oxaliplatin; KP 1339

STUDY DESIGN:
Intervention Model Description: Randomized - Arm VII only: Second line mCRC 500 mg/m2 or 625 mg/m2 in combination with FOLFOX or FOLFOX alone, in a 1:1:1 ratio.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Part B - Dose Expansion - 1L Gastric Cancer (ARM I) (Experimental): Arm closed to enrollment.
  Interventions: Drug: BOLD-100 in combination with FOLFOX Chemotherapy (Arms I-VI)
- Part B - Dose Expansion - 2L Gastric Cancer (ARM II) (Experimental): Arm closed to enrollment.
  Interventions: Drug: BOLD-100 in combination with FOLFOX Chemotherapy (Arms I-VI)
- Part B - Dose Expansion - 2L Pancreatic Cancer (ARM III) (Experimental): Arm closed to enrollment.
  Interventions: Drug: BOLD-100 in combination with FOLFOX Chemotherapy (Arms I-VI)
- Part B - Dose Expansion - 2L Colorectal Cancer (ARM IV) (Experimental): Arm closed to enrollment.
  Interventions: Drug: BOLD-100 in combination with FOLFOX Chemotherapy (Arms I-VI)
- Part B - Dose Expansion - 2L Cholangiocarcinoma (ARM V) (Experimental): Arm closed to enrollment.
  Interventions: Drug: BOLD-100 in combination with FOLFOX Chemotherapy (Arms I-VI)
- Part B - Dose Expansion - 3L Colorectal Cancer (ARM VI) (Experimental): Arm closed to enrollment.
  Interventions: Drug: BOLD-100 in combination with FOLFOX Chemotherapy (Arms I-VI)
- Part B - Dose Expansion - 2L Colorectal Cancer (ARM VIIA) (Active Comparator): Arm open to enrollment. 500 mg/m2 BOLD-100 + SOC FOLFOX
  Interventions: Drug: BOLD-100 +/- FOLFOX Chemotherapy (Arm VII)
- Part B - Dose Expansion - 2L Colorectal Cancer (ARM VIIB) (Active Comparator): Arm open to enrollment. 625 mg/m2 BOLD-100 + FOLFOX
  Interventions: Drug: BOLD-100 +/- FOLFOX Chemotherapy (Arm VII)
- Part B - Dose Expansion - 2L Colorectal Cancer (ARM VIIC) (Active Comparator): Arm open to enrollment. FOLFOX alone.
  Interventions: Drug: BOLD-100 +/- FOLFOX Chemotherapy (Arm VII)

INTERVENTIONS:
Drug: BOLD-100 +/- FOLFOX Chemotherapy (Arm VII) — Arm VIIA: 500 mg/m2 BOLD-100 combined with FOLFOX; Arm VIIB: 625 mg/m2 BOLD-100 combined with FOLFOX; Arm VIIC: FOLFOX alone
  Other Names: BOLD-100 +/- Folinic acid (leucovorin), Fluorouracil (5-FU), and Oxaliplatin.
  Arms: Part B - Dose Expansion - 2L Colorectal Cancer (ARM VIIA); Part B - Dose Expansion - 2L Colorectal Cancer (ARM VIIB); Part B - Dose Expansion - 2L Colorectal Cancer (ARM VIIC)
Drug: BOLD-100 in combination with FOLFOX Chemotherapy (Arms I-VI) — BOLD-100 at 625 mg/m2 combined with FOLFOX Chemotherapy
  Other Names: BOLD-100 +/- Folinic acid (leucovorin), Fluorouracil (5-FU), and Oxaliplatin.
  Arms: Part B - Dose Expansion - 1L Gastric Cancer (ARM I); Part B - Dose Expansion - 2L Cholangiocarcinoma (ARM V); Part B - Dose Expansion - 2L Colorectal Cancer (ARM IV); Part B - Dose Expansion - 2L Gastric Cancer (ARM II); Part B - Dose Expansion - 2L Pancreatic Cancer (ARM III); Part B - Dose Expansion - 3L Colorectal Cancer (ARM VI)

SUMMARY:
BOLD-100 is an intravenously administered sterile solution containing the ruthenium-based small molecule. BOLD-100 has been shown to preferentially decrease the expression of GRP78 in tumour cells and ER stressed cells when compared to normal cells. BOLD-100 will be combined with cytotoxic FOLFOX chemotherapy in this study, with a dose escalation cohort to ensure tolerability and safety, followed by a cohort expansion phase.

DETAILED DESCRIPTION:
BOLD-100 is a novel, targeted anti-cancer therapy which is an intravenously administered small molecule drug. In a previous Phase 1 study (NCT01415297) BOLD-100 showed low toxicity with minimal hematological issues as well as some potential anti-tumour activity. The lack of observed hematological toxicity and neurotoxicity position BOLD-100 well for use in combination with a broad range of standard-of-care (SOC) chemotherapy regimens.

This is a prospective, multicenter non-randomized Phase 1b/2a dose escalation & expanded cohort study of BOLD-100 in patients with advanced gastrointestinal malignancies (colorectal, pancreatic, gastric cancers, and cholangiocarcinoma) receiving standard-of-care FOLFOX chemotherapy. Enrollment in Arms I - VI is closed to enrollment.

Colorectal cancer (ARM VII) for patients who are oxaliplatin naïve and have received only 1 prior line of therapy in the metastatic setting. Within this arm, participants will be randomized to one of two dose levels of BOLD-100 - either 500 mg/m2 or 625 mg/m2 in combination with FOLFOX or FOLFOX alone, in a 1:1:1 ratio. Participants enrolled into Arm VII will complete quality of life questionnaires examining general quality of life and neuropathy associated quality of life parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 years or older.
2. Be male or non-pregnant females who agree to comply with applicable contraceptive requirements of the protocol.
3. Histologically and/or cytologically confirmed gastrointestinal tumours that are metastatic or unresectable. (ARM VII): Patients must have received only 1 prior line of therapy in the metastatic setting.
4. Have measurable disease according to RECIST v1.1.
5. Have an anticipated survival of at least 16 weeks.
6. Be ambulatory, with an ECOG performance score of 0 or 1.
7. Have adequate organ function.
8. Be on stable doses of any drugs that may affect hepatic drug metabolism or renal drug excretion.
9. Be fully informed about their illness and the investigational nature of the study protocol, and sign a REB-approved Informed Consent Form (ICF).
10. (ARM VII): BRAF wild-type tumour status.

Exclusion Criteria:

1. Neuropathy > grade 2
2. Previous intolerance to or significant reaction secondary to fluorouracil or oxaliplatin.
3. Cerebrovascular accident within the past 6 months before the start of treatment.
4. History or presence of central nervous system (CNS) metastasis or leptomeningeal tumours.
5. Any serious medical conditions that might be aggravated by treatment or limit compliance.
6. Any history of serious cardiac illness.
7. Hemoptysis, cerebral, or clinically significant gastrointestinal hemorrhage in the past 6 months before the start of treatment.
8. Any other known malignancy within 3 years before the start of treatment.
9. Active gastrointestinal tract disease with malabsorption syndrome.
10. Non-healing wound, fracture, or ulcer, or presence of symptomatic peripheral vascular disease.
11. Treatment with radiation therapy or surgery within 4 weeks prior to starting treatment.
12. Recent history of weight loss > 10% of current body weight in past 3 months before the start of treatment.
13. HIV-positive subjects on combination anti-retroviral therapy due to the potential for PK interactions with the study agent.
14. Concurrent use of another investigational therapy or anti-cancer therapy within 4 weeks before the start of treatment.
15. Currently breastfeeding
16. Dihydropyrimidine Dehydrogenase (DPD) deficiency
17. Current or prior treatment with potent inhibitors of Dihydropyrimidine Dehydrogenase (DPD)
18. (ARM VII): Prior exposure to BOLD-100
19. (ARM VII): Subjects with microsatellite-high (MSI-H) Tumours
20. (ARM VII): Concurrent monoclonal antibody therapy for mCRC (anti-EGFR, anti-VEGF or anti-HER2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2020-08-28 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events ([S]AEs) | Through study completion, approximately 2 weeks after last treatment
  Arms I-VI: Primary outcome measure; Arm VII: Secondary outcome measure
Incidence of dose-limiting toxicities (DLT) | Screening to 4 weeks after first treatment
  Dose escalation only.
Incidence of clinically significant changes or abnormalities from Physical Examinations, ECGs, Vital Signs, Laboratory Results, ECOG performance status | Through study completion, approximately 2 weeks after last treatment
  Arms I-VI: Primary outcome measure; Arm VII: Secondary outcome measure
Progression Free Survival (PFS): Arm VII | Through study completion, approximately 2 weeks after last treatment for last patient
  Arm VII: Primary outcome measure
Overall Response Rate (ORR): Arm VII | Through study completion, approximately 2 weeks after last treatment for last patient
  Arm VII: Primary outcome measure
Overall Survival (OS): Arm VII | Through study completion, approximately 2 weeks after last treatment for last patient
  Arm VII: Primary outcome measure

SECONDARY OUTCOMES:
Progression Free Survival (PFS): Arms I-VI | Through study completion, approximately 2 weeks after last treatment for last patient
  Arms I-VI: Secondary outcome measure
Overall Response Rate (ORR): Arms I-VI | Through study completion, approximately 2 weeks after last treatment for last patient
  Arms I-VI: Secondary outcome measure
Overall Survival (OS): Arms I-VI | Through study completion, approximately 2 weeks after last treatment for last patient
  Arms I-VI: Secondary outcome measure
Baseline and changes in biomarker levels during treatment | Arms I-VII; Through study completion, approximately 2 weeks after last treatment
  Serum GRP78
Peak Plasma Concentrations (Cmax) | Arms I-VII; Through study completion, approximately 2 weeks after last treatment
  Arms I-VII
Area under the plasma concentration versus time (AUC) | Arms I-VII; Through study completion, approximately 2 weeks after last treatment
  Arms I-VII
Elimination half life (T1/2) | Arms I-VII; Through study completion, approximately 2 weeks after last treatment
  Arms I-VII

OTHER OUTCOMES:
Quality of life evaluation | Through study completion, approximately 2 weeks after last treatment
  Arm VII
Changes in dose reductions, treatment discontinuations, and interruptions, and AE's reported related to neuropathy from baseline | Through study completion, approximately 2 weeks after last treatment
  Arm VII
Cancer mutational status in blood and tissue biomarker relationship to clinical outcomes | Arm VII; Through study completion, approximately 2 weeks after last treatment
  Circulatory tumor DNA (ctDNA) collection will be tested for a panel of tumor mutations, genomic alterations, microsatellite instability and tumor mutational burden, and these will be associated to clinical outcomes, including overall survival, progression-free survival, overall response rate and other outcome measures
GRP78 levels and relationship to clinical outcomes | Arm VII; Through study completion, approximately 2 weeks after last treatment
  Optional biopsy samples at screening and at cycle 4 will be collected and analyzed for GRP78 levels, other related pathway markers, immune cell profiles, and cancer mutation profiles, and comparing these to clinical outcomes including overall survival, progression-free survival, overall response rate and other outcome measures

CONTACTS AND LOCATIONS:
Locations (16):
- United States (2):
  - University of California, Los Angeles, Santa Monica, California
  - Moffitt Cancer Center, Tampa, Florida
- Canada (6):
  - Cross Cancer Institue, Edmonton, Alberta
  - Juravinski Cancer Centre, Hamilton, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre Glen Site, Montreal, Quebec
- Ireland (3):
  - Mater Miserecordiae University Hospital, Dublin
  - St. James Hospital, Dublin
  - St. Vincent's University Hospital, Dublin
- South Korea (5):
  - National Cancer Center, Goyang
  - Kangbuk Samsung Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital - Yonsei University, Seoul

IPD SHARING:
Plan to Share IPD: No